CLINICAL TRIAL: NCT06897488
Title: EMERALD: Endocrine Therapy oMission With Radiation in ER+ Breast Cancer: Assessing Quality of Life and Disease Control: a Prospective Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0191; NCI-2025-02147 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-03-25; First posted 2025-03-27 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endocrine Therapy (Experimental)
  Interventions: Radiation: Adjuvant Radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Participants will receive treatment following Lumpectomy

SUMMARY:
This clinical research study is to learn about the effects of giving radiotherapy alone after lumpectomy to patients who have early-stage, low-risk breast cancers and who are 60 years of age or older.

DETAILED DESCRIPTION:
Primary Objective:

To determine the 3- year DMFS rate of radiotherapy as adjuvant monotherapy for early stage, low risk breast cancers in patients aged ≥ 60 years

Secondary Objectives:

1. To determine the HRQoL of patients ≥ 60 years with early stage, low risk breast cancer receiving adjuvant monotherapy with radiotherapy
2. To determine the 3-year and 5-year risk of ipsilateral breast tumor recurrence (IBTR) for early-stage breast cancers treated with lumpectomy and adjuvant radiotherapy without endocrine therapy
3. To quantify the 3-year and 5-year rates of local-regional recurrence, contralateral breast cancer, breast cancer-specific survival and overall survival and the 5 year rate of DMFS
4. To determine the 5-year utilization of salvage mastectomy and other salvage therapies
5. To determine late (up to 11 year) oncologic outcome data for patients accessible via chart review or phone call
6. To determine the toxicities experienced by patients ≥ 60 years with early stage, low risk breast cancer receiving adjuvant monotherapy with radiotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pathologically-confirmed invasive breast cancer
2. Age ≥ 60 years
3. Treatment with breast conserving surgery
4. Pathologic T stage of T1 or T2 with total tumor size ≤ 3cm including any component of DCIS that may exist in conjunction with invasive disease
5. Ki-67 . 20% and/or Oncotype 0-10 (Ultra Low)
6. Final surgical margins negative, defined as no tumor on ink. Lobular carcinoma in situ involving the final surgical margin will be disregarded.
7. Tumor must be estrogen receptor positive, progesterone receptor positive and HER2Neu non-amplified as per current College of American Pathologists guidelines
8. Clinical nodal stage cN0
9. If pathologic nodal staging is obtained, then pN0 or pN0(i+)
10. Patients have had or have a scheduled discussion with a breast medical oncologist regarding adjuvant treatment options
11. Patients who have met criteria 4.1.1-4.1.9 who never initiate endocrine therapy OR who initiate adjuvant endocrine therapy but discontinue it within 6 months of initiation * In some clinical scenarios, patients may have a particularly small volume of tumor, making it not be feasible for all of these biomarkers to be evaluated. In this scenario, if the PI and/or Protocol Collaborators are able to document that a patient is being treated as if they have luminal A (biologically favorable) breast cancer then the patient is eligible for enrollment if all other eligibility criteria are met.

Exclusion Criteria:

1. Node positive disease (N1-3)
2. Metastatic disease (M1)
3. Grade 3 disease and lymphovascular space invasion in the tumor
4. Synchronous bilateral breast cancer
5. Receipt of neoadjuvant therapy
6. Diagnosis of a collagen vascular disease associated with an increased incidence of radiation toxicities such as scleroderma or systemic lupus erythematosis
7. Diagnosis of other cancer within the prior 5 years, excluding basal or squamous cell carcinoma of the skin that has been treated
8. Patient with psychiatric illness/social situations that would limit compliance with study requirements
9. Prior radiotherapy to the index breast or recurrent cancer of the breast
10. Known carrier of a mutation associated with predisposition to breast cancer development, including BRCA1 or BRCA2

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 300 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Simona Shatelman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org